CLINICAL TRIAL: NCT05780892
Title: A Randomized-Controlled Trial to Reduce Clinician Burnout
Brief Title: Keck Medicine of University of Southern California Thrive Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Steven Siegel, Professor of Psychiatry, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UniHealth Foundation 5125
Record Dates: First submitted 2023-03-10; First posted 2023-03-23 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Burnout
Keywords: healthcare worker; clinician; wellness; process improvement; electronic health record
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial of 3 interventions for clinician well-being as compared to controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Emotional Wellbeing (Experimental): This arm consists of 6 30-minute group sessions taking place every 2 weeks for a total of 12 weeks. The sessions will be led by licensed therapists based on cognitive behavioral therapy and acceptance and commitment therapy. Session topics are sequential in nature such that each session builds on the previous session. Between sessions, participants will complete worksheets based on the material covered in the previous session. If a participant misses a session, they will be provided with a pre-recording with the content they missed.
  Interventions: Behavioral: Emotional Wellbeing
- EHR Skills Optimization (Experimental): This arm consists of 6 individual educational sessions taking place every 2 weeks for a total of 12 weeks which will be scheduled to accommodate clinicians schedule and preferences. These sessions will be led by a member of the clinical informatics team and target optimization of the EHR. The sessions will be conducted on site, virtually, or a combination of both onsite and virtual. Between sessions participants are to note any challenges, questions, or recommendations related to the EHR. If participant misses 2 sessions, they will be asked to reschedule, but if they miss 3 sessions they may be asked to withdraw from the intervention.
  Interventions: Behavioral: EHR Skills Optimization
- Performance Improvement (Experimental): This arm consists of 6 virtual group sessions taking place over every 2 weeks for a total of 12 weeks. The sessions target improving perceptions of the work environment through foundational performance improvement knowledge and skills, and they will be led by a member of the systems-reengineering team. Between sessions, participants will be asked to follow through on tasks outlined in the learning sessions and share in the next session. If a session is missed, they will be provided with a prerecording of the didactic material presented in the learning sessions.
  Interventions: Behavioral: Performance Improvement
- Control (Active Comparator): Participants randomly assigned to the control condition will continue as usual care and will not complete any intervention during the duration of the study.
  Interventions: Behavioral: control

INTERVENTIONS:
Behavioral: Emotional Wellbeing — Participants in this intervention will learn cognitive behavioral therapy tools to identify unhelpful beliefs and thought patterns, increase motivation through SMART goal making, and increase relaxation and stress management techniques through deep breathing, progressive muscle relaxation and pleasant activity scheduling. Additionally, participants will learn acceptance and commitment therapy tools to increase cognitive flexibility and resilience through acceptance and diffusion work, being present through contact with present moment and self as context and doing what matters through committed actions and value identification.
  Arms: Emotional Wellbeing
Behavioral: EHR Skills Optimization — Participants in this intervention will learn how to better utilize the EHR by gaining knowledge and skills in the EHR. Session topics include, but are not limited to, understanding current usage patterns and behaviors in the EHR, optimization of the table of contents for easier chart navigation, integration of specialty-focused workflows with current EHR documentation and chart review tools, and recommendations to be more efficient and reduce amount of time spent in the EHR.
  Arms: EHR Skills Optimization
Behavioral: Performance Improvement — This intervention focuses on improving participants perception of Keck Medicine as a positive workplace environment by supporting participants in gaining basic performance improvement knowledge and skills through didactic training, group discussions based on sociocultural learning theory, and hands on practice leading a performance improvement project. Sessions will review performance improvement concepts such as Lean wastes, systems thinking, change management and sustainability. Participants in this intervention will then identify a project area of focus that they want to improve and develop a project charter. Once a project area has been identified, participants will be put into breakout rooms to discuss successes and challenges as well as receive feedback on their project from peers.
  Arms: Performance Improvement
Behavioral: control — Participants randomly assigned to the control condition will continue as usual care and will not complete any intervention during the duration of the study.
  Arms: Control

SUMMARY:
Burnout and job dissatisfaction among clinicians are one of the greatest challenges facing healthcare today. Clinicians report feeling less engaged in their work and are leaving their fields in large numbers which reflects increasing stress from the pandemic coupled with increased administrative and regulatory demands and a decreased sense of autonomy. To attenuate these factors the current study will enact a series of interventions that would decrease mental distress, increase self-efficacy, and attenuate inefficiencies in their work environment to achieve sustainable improvement. The investigators will offer psychological training using techniques that have been shown to impact individual's mental health that target feelings of demoralization, depression and anxiety that result from chronic stress. Additionally, the investigators will offer individualized training on optimization of the Electronic Health Record (EHR) to help clinicians from different fields and settings reduce their time and effort needed for documentation. The investigators will also engage clinicians in systemic redesign to empower clinician-directed changes to the health system environment. The investigators anticipate that each intervention will positively affect emotional wellbeing, skills mastery of the Electronic Health Record (EHR), and environmental dissatisfaction to reduce overall burnout.

DETAILED DESCRIPTION:
This study is a randomized controlled trial to reduce burnout that is frequently experienced among clinicians. Personal burnout can be defined as a state of emotional, physical, and mental exhaustion created by excessive and prolonged stress occurring when one feels overwhelmed, emotionally drained, and unable to meet constant demands. The need to improve clinician burnout is higher than ever before due to increased intensity and duration of chronic stress resulting from the COVID-19 pandemic. However, there are significant barriers to attenuating burnout experienced by clinicians, some of which are extrinsic such as the severe nature of the COVID-19 pandemic, and some are intrinsic such as pressure of increased productivity. Previous research has focused on increasing clinician wellness through improving their toleration of difficulties in the work environment and has concluded that no single intervention is effective in promoting and maintaining wellbeing but utilizing multiple interventions could have an additive effect. The goal of the current study is to determine the extent to which different interventions impact clinician burnout. Each intervention in this study targets a unique aspect of burnout including emotional wellbeing, skill using the Electronic Health Record (EHR), and factors that contribute to dissatisfaction in the workplace. The results from this study will guide future programs to reduce burnout at Keck Medicine and the broader health environment.

Clinicians cannot effectively function in their jobs if they feel overwhelmed, depressed, or anxious, so the investigators will address the emotional state of clinicians using Cognitive Behavioral Therapy (CBT) and Acceptance and Commitment Therapy (ACT) to reduce measures of depression and anxiety while increasing measures of resilience. The investigators anticipate that learning how to employ the principles of Cognitive Behavioral Therapy (CBT) and Acceptance and Commitment Therapy (ACT) will result in improvements in clinicians' emotional wellbeing. This intervention will consist of training sessions led by licensed therapist and will utilize Cognitive Behavioral Therapy-based skills, such as cognitive restructuring to identify unhelpful behaviors and thought patterns, relaxation strategies such as deep breathing, and acceptance and commitment therapy-based skills such as increasing psychological flexibility. Participants in this intervention group will complete the Patient General Health Questionnaire (PHQ-9) and Brief Resilience Scale (BRS) prior to the intervention, immediately following the intervention, and 6 months after completion of the intervention. These scores will be compared to the scores of the control group to determine the impact of this intervention.

Additionally, if clinicians lack mastery of key skills needed to do their jobs quickly and efficiently they are likely to feel overwhelmed and overworked. Self-efficacy beliefs will be addressed by teaching clinicians how to better use the Electronic Health Record (EHR) to reduce frustrations at work and time spent in the EHR, increase percentage of clinical notes completed on time, and decrease the need to revise clinical records. Augmented specialty and site-specific training will be provided to improve current capabilities in the EHR and identify areas for improvement in EHR configuration. Preintervention data will also be collected and shared with study participants which includes but is not limited to actual EHR per patient, time spent in EHR after hours, and chart review time per patient. The investigators anticipate that learning how to better use the EHR for one's field and setting will increase scores for self-efficacy and reduced frustrations at work. To assess the immediate and long-term impact of the intervention, participants in this intervention will complete a newly developed survey by the study team pertaining to participant's skills and satisfaction with the EHR system prior to the intervention, immediately following the intervention and 6 months after the intervention.

Perceptions of a poor work environment such as too much workload, low control or being treated unfairly will negatively impact clinicians' ability to do their job and remain engaged in their field. This dissatisfaction will be addressed by providing participants with basic performance improvement knowledge and skills through didactic training, group discussions, and hands on practice leading a performance improvement project. The performance improvement concepts are Lean, systems thinking, change management and sustainability. To assess the immediate and long-term impact of this intervention, participants will complete a modified version of the Beliefs, Attitudes, Skills and Confidence in Quality Improvement (BASiC-QI) scale prior to the intervention, immediately following the intervention, and 6 months after the intervention. The investigators anticipate that participating in systemic redesign will increase participants perception of Keck Medicine as a positive work environment and this environmental improvement will have collateral benefit for a reduction in clinician departures.

In addition to the 3 interventions, there will also be a control condition in which the participants do not complete any intervention to control for impact of changes in their lives, subsequent pandemic variants, or other world stressors on evaluations of mental state. The control participants will complete the same assessments at the same time points as the intervention participants. The assessment scores of the participants in each intervention condition will be compared to the scores of participants in the control condition allowing the investigators to study the impact of the different interventions.

Statistical analyses will focus on examining whether participation in the interventions leads to reductions in burnout, improvement in wellbeing, and greater work efficiency and job satisfaction immediately after treatment and at 6-month follow-up. Data will be assessed in accordance with the intent to treat (ITT) principle for all primary analyses on treatment effects. The investigators will use repeated measure analyses of covariance models. The investigators will first conduct an omnibus test for both post treatment assessment periods to examine the overall effect of each intervention followed by separate tests for each posttreatment assessment period of the study. Estimated intervention effects will be derived as the group difference in change from baseline to a specific assessment period. Intervention effect sizes will be calculated with Cohen's d and standardized response mean as the group difference in change relative to the SD of change scores. Additionally, the Wellbeing Index will be evaluated across all active arms compared to a control using an ANOVA with study arms as the independent variables such that the investigators can then look for an interaction between active arms and outcomes enabling the investigators to look at each arm individually.

ELIGIBILITY:
Inclusion Criteria:

Credentialed providers (e.g., MD/PA/NP across all specialties or clinical Ph.D./MS) or direct care providers/clinicians (e.g., RN, LVN, OT, PT, SLP, RT) within the Keck Medical System.

Exclusion Criteria:

a. Non-faculty or non-clinical staff (e.g., residents, administrators, etc.) at Keck Medicine

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in emotional well-being | Participants will complete this survey at baseline, immediately following the intervention, and 6 months after completion of the intervention.
  Emotional wellbeing will be assessed by a change in baseline on the Patient Health Questionnaire (PHQ-9) which is a 9-item validated survey designed to measure symptoms of depression. This scale incorporates the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria into self-reported scores of wellbeing. Responses are on a 0-3 scale based on frequency of symptoms. A score of 0 corresponds to "not at all" and a score of 3 corresponds to "nearly every day."
Change in Resilience | Participants will complete this survey at baseline, immediately following the intervention, and 6 months after completion of the intervention
  Resilience will be assessed by a change in baseline on the Brief Resilience Scale (BRS) which is a 6-item validated scale measuring a participant's perception of their ability to bounce back from stressful events. The responses are on a 5-point Likert scale based on extent of agreement with the statements on the scale. Statements 1,3, and 5 are positively worded and statements 2,4, and 6 are negatively worded, so responses are scored by reverse coding statements 2,4, and 6. A score of 1 corresponds to "Strongly Disagree" and a score of 5 corresponds to "Strongly Agree".
Change in EHR Skills and Optimization | Participants will complete this survey at baseline, immediately following the intervention, and 6 months after completion of the intervention.
  EHR Skills and optimization will be assessed using a newly developed 7-item survey by the study team that pertain to an individual's skills and satisfaction with the EHR. Responses are on a 5-point Likert scale based on extent of agreement with the statements on the scale. A score of 1 corresponds to "Strongly Disagree" and a score of 5 corresponds to "Strongly Agree."
Change in Electronic Health Record (EHR) Proficiency | Participants will complete this survey at baseline, immediately following the intervention, and 6 months after completion of the intervention.
  Objective measures of EHR proficiency will include percentage of clinical notes completed on time, reduction in time spent using the EHR and reduction in need to revise clinical records among study participants in the EMR skills acquisition group. These will be compared to the same measures among study participants in other arms of this study, as well as system wide trends for all measures over the study interval.
Change in perceptions of Quality Improvement | Participants will complete this survey at baseline, immediately following the intervention, and 6 months after completion of the intervention
  Perceptions of Quality/Performance Improvement will be assessed by a change in baseline scores on the Beliefs, Attitudes, Skills, and Confidence in Quality Improvement (BASiC-QI) Scale. The BASiC-QI Scale is 31-item multidimensional self-assessment to assess knowledge, skills, and attitudes about Quality Improvement. The statements in the survey are in sequential order by which one would design a QI project. The responses for the beliefs and attitudes subscale and the knowledge subscale are on a 7-point Likert scale based on extent of agreement with the statements. A score of 1 corresponds to "Strongly Disagree" and a score of 7 corresponds to "Strongly Agree". The QI Skills subscale responses are a continuum of confidence level about the statements, with a score of 1 corresponding to "Not confident whatsoever" and a score of 4 corresponds to "Extremely Confident."
Change in score of Proficiency improvement | Participants will complete this survey at baseline, immediately following the intervention, and 6 months after completion of the intervention
  NIH Proficiency Scale assesses, "How would you rate your level of expertise?" using the following options:
  1. Fundamental Awareness (basic knowledge)
  2. Novice (limited experience)
  3. Intermediate (practical application)
  4. Advanced (applied theory)
  5. Expert (recognized authority)
Change in Environmental Satisfaction | Participants will complete this survey at baseline, immediately following the intervention, and 6 months after completion of the intervention.
  Environmental satisfaction will be assessed using the Safety, Culture, Operational Risk, Resilience/Burnout and Engagement (SCORE) survey. The SCORE survey is an outcomes-predictive and proprietary established scale designed to measure satisfaction in the workplace. The responses are based on extent of agreement with the statements. A score of 1 corresponds to "Strongly Disagree", a score of 5 corresponds to "Strongly Agree", and a score of 6 corresponds to "not applicable."
Change in Burnout | Participants will complete this survey at baseline, immediately following the intervention, and 6 months after completion of the intervention.
  Burnout levels will be assessed using the 7- item Personal Burnout subscale of the SCORE survey. The responses are based on extent of agreement with the statements. A score of 1 corresponds to "Strongly Disagree", a score of 5 corresponds to "Strongly Agree", and a score of 6 corresponds to "not applicable."
Change in Overall Well-being | Participants will complete this survey at baseline, immediately following the intervention, and 6 months after completion of the intervention.
  Overall well-being will be assessed using the 7-item Wellbeing Index. The Well-being Index identifies distress in a variety of dimensions such as anxiety and fatigue. The response choices are either "yes" or "no" based on whether the participant has experienced the symptoms described in the scale.

SECONDARY OUTCOMES:
Change in Emotional Thriving | : participants will complete this survey at baseline, immediately following the intervention, and 6 months after completion of the intervention
  Emotional Thriving will be assessed using the 5-item Emotional Thriving Subscale of the SCORE Survey. The responses are based on extent of agreement with the statements. A score of 1 corresponds to "Strongly Disagree", a score of 5 corresponds to "Strongly Agree", and a score of 6 corresponds to "not applicable."
Change in Emotional Recovery | participants will complete this survey at baseline, immediately following the intervention, and 6 months after completion of the intervention
  Emotional Recovery will be assessed using the 4-item Emotional Recovery subscale of the SCORE Survey. The responses are based on extent of agreement with the statements. A score of 1 corresponds to "Strongly Disagree", a score of 5 corresponds to "Strongly Agree", and a score of 6 corresponds to "not applicable."
Change in Workload | participants will complete this survey at baseline, immediately following the intervention, and 6 months after completion of the intervention
  Perceptions of workload will be assessed using the 7-item Workload Subscale of the SCORE Survey which identifies the demands that contribute ti a workload that is increasingly demanding and stressful to manage. The responses are based on extent of agreement with the statements. A score of 1 corresponds to "Strongly Disagree", a score of 5 corresponds to "Strongly Agree", and a score of 6 corresponds to "not applicable."
Change in Intent to Leave | participants will complete this survey at baseline, immediately following the intervention, and 6 months after completion of the intervention
  Participant's intent to leave will be assessed using the 3-item Intent to Leave subscale of the SCORE Survey. The responses are based on extent of agreement with the statements. A score of 1 corresponds to "Strongly Disagree", a score of 5 corresponds to "Strongly Agree", and a score of 6 corresponds to "not applicable."
Change in Participation in Decision Making | participants will complete this survey at baseline, immediately following the intervention, and 6 months after completion of the intervention
  The Participation in Decision-Making will be assessed using the 6-item Participation in Decision-Making subscale of the SCORE survey which evaluates the current state of the decision-making process and participant's perception of their level of participation in the decision-making process. The responses are based on extent of agreement with the statements. A score of 1 corresponds to "Strongly Disagree", a score of 5 corresponds to "Strongly Agree", and a score of 6 corresponds to "not applicable."

CONTACTS AND LOCATIONS:
Overall Officials: Steven Siegel, MDPhD, Principal Investigator — University of Southern California
Locations (1):
- Keck School of Medicine, University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruple C, Brodhead J, Rabinovich L, Junghaenel DU, Nakamura T, Wong J, De-Oliveira S, Brown J, Nguyen P, Horn J, Middleton R, Brahe M, Wen C, Rao S, Nguyen C, Shlamovitz G, Marino D, Osorno F, Siegel S. Protocol of randomized-controlled trial to examine the effectiveness of three different interventions to reduce healthcare provider burnout. BMC Health Serv Res. 2024 Dec 23;24(1):1643. doi: 10.1186/s12913-024-12131-4. PMID 39716202